CLINICAL TRIAL: NCT07188519
Title: A Study of Effects of Expressive Writing on College Students Experiencing Psychological Difficulties
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Siwei Zhu, Dr, Shandong University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ECSBMSSDU2023-1-85
Record Dates: First submitted 2025-09-16; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Negative Emotions; Self Cognition

STUDY DESIGN:
Intervention Model Description: The intervention with EW on Anne followed the design of Pennebaker and Beall (1986) with adjusted writing tasks based on Tolcher et al. (2024) (See Figure 1). Lasting for 40 days, it included four rounds of writing with a detached vantage point-one month, three months, and six months after the intervention Each of the four rounds consisted of three consecutive days of writing followed by a gap week. On each day, Anne was asked to write continuously for 20-25 minutes about her life experiences that had a significant impact on her, either positively or negatively. After writing on the third day of each round, Ann responded to the BDI-II and answered interview questions about her emotional state and self-cognition. The gap week was intended to facilitate her psychological adjustment and prevent emotional overwhelm and habituation. It is an important component of the healing process, allowing for the deep, unconscious work of integration, meaning-making, and emotional regulation to occur.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- case study (Other): The intervention with EW on participants followed the design of Pennebaker and Beall (1986) with adjusted writing tasks based on Tolcher et al. (2024). Lasting for 40 days, it included four rounds of writing with a detached vantage point-one month, three months, and six months after the intervention Each of the four rounds consisted of three consecutive days of writing followed by a gap week. On each day, they were asked to write continuously for 20-25 minutes about her life experiences that had a significant impact on her, either positively or negatively. After writing on the third day of each round, they responded to the BDI-II and answered interview questions about their emotional state and self-cognition.
  Interventions: Other: expressive writing

INTERVENTIONS:
Other: expressive writing — Each of the four rounds consisted of three consecutive days of writing followed by a gap week.

SUMMARY:
This study aims to improve college students' mental health through expressive writing. Over the next eight weeks, I would like you to write about some of the experiences that have had the greatest impact on your life. These may be positive or negative, and may relate to the present, past, or future. As you write, you may describe the event from both positive and negative perspectives. We encourage you to genuinely explore your deepest emotions and thoughts. Whatever you choose to write about, the crucial point is that you truly delve into your innermost feelings and reflections. You may relate your experiences to anyone in your life, including your parents, friends, and relatives. We hope you will endeavour to write about significant experiences you have never discussed in detail with others. During your writing, do not concern yourself with linguistic expression. We wish for you to convey your deepest emotions and thoughts as fully as possible. The content of your writing will not influence our perception of you; it is held in absolute confidence and security. The sole rule for this writing session is that once you begin writing, you must continue until the time concludes (each session is timed for 20-25 minutes). After the writing period ends, you may choose whether to submit your written text.

ELIGIBILITY:
Inclusion Criteria:

1. A score indicating mild or higher depressive symptoms on the Beck Depression Inventory (BDI);
2. Age ranging from 18 to 29 years old;
3. Educational background of undergraduate degree or above; -

Exclusion Criteria:

1. Participants with no depressive symptoms
2. Participants with writing difficulties, dysgraphia, or dyslexia
3. Participants with severe physical illnesses or without civil capacity -

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2023-11-02 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
self cognition | From enrollment to the end of study at one year.
  Additionally, to assess changes at cognitive levels, we separately recorded and compared the items related to self-cognition (7 items) within the BDI-II. The specific determination rules were as follows:the direction of score change at the item level served as the basis for judgement. Within a given assessment interval, we compared the number of items that decreased (indicating improvement) with those that increased (indicating deterioration). If decreases outnumbered increases, we classified the interval as improvement-predominant; otherwise, deterioration predominated. If the two were comparable, the change was recorded as insignificant. Accordingly, we sequentially compared items across the self cognition dimensions in the nine assessments, thereby revealing the immediate and sustained manifestations of expressive writing at both cognitive levels. Besides, the cognitive words and self cognition related sentences in interview were also analysis as the evidences for self cognition.
negative emotion and positive emotion | From enrollment to the end of study at one year
  we separately recorded and compared the items related to emotional state (5 items) The specific determination rules were as follows: the direction of score change at the item level served as the basis for judgement. Within a given assessment interval, we compared the number of items that decreased (indicating improvement) with those that increased (indicating deterioration). If decreases outnumbered increases, we classified the interval as improvement-predominant; otherwise, deterioration predominated. If the two were comparable, the change was recorded as insignificant. Accordingly, we sequentially compared items across the negtaive emotion and positive emotion dimensions in the nine assessments, thereby revealing the immediate and sustained manifestations of expressive writing at both emotional levels. Besides, the emotional words used in the writing texts and emotional related senteneces in semi-strcutured interview also analysis as the evidences for positive and negtaive emotion.

CONTACTS AND LOCATIONS:
Locations (1):
- Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided
The datasets generated and analyzed during the current study contain potentially identifiable information about research participants. As explicit consent for public data release was not obtained from participants, the raw data cannot be made publicly available to protect their privacy. Requests for access to de-identified data (where permissible) may be directed to the corresponding author and will be reviewed on a case-by-case basis in accordance with ethical guidelines